CLINICAL TRIAL: NCT05514977
Title: Ultrasound Guided Thoracic Erector Spine Plane Block for Post Mastectomy Pain Control, Effect of Volume With Constant Drug Mass, a Randomized Controlled Trial
Brief Title: Ultrasound Guided Thoracic ESPB for Post Mastectomy Pain Control, Comparing 2 Dosing Regimens of Lidocaine With Different Drug Volumes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kareem, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LOW VS HIGH VOLUME LIDOCAINE
Record Dates: First submitted 2022-05-19; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L group (Active Comparator): Patients are given 20 ml of 2 % lidocaine for ESPB
  Interventions: Procedure: Erector spine plane block
- H group (Active Comparator): Patients are given 40 ml of 1 % lidocaine for ESPB
  Interventions: Procedure: Erector spine plane block

INTERVENTIONS:
Procedure: Erector spine plane block — Thoracic ESPB

SUMMARY:
The investigators compare 2 different drug regimens using 2 different volumes of lidocaine with the same drug content (i.e. different concentrations) as regards efficacy of post operative analgesia following mastectomy surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA 2 & 3 for elective breast cancer surgery

Exclusion Criteria:

* ASA > 3
* BMI > 35 kg/m2
* Contraindications to LA (coagulopathy and local infection)
* Allergy to the drug
* Cardiac, hepatic and renal patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Effective analgesia | First 24 hours
  Morphine supplements needed

SECONDARY OUTCOMES:
Analgesic efficiency | Every 2 hours in the first 24 hours
  Visual analog scale; ranging from 0 to 10 where 0 is no pain and 10 is pain in its worst form

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kareem, Study Director — Kasr alainy hospital, Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No